CLINICAL TRIAL: NCT04924556
Title: The Effect of Rıgıd Brace on Spinopelvic Parameters and GAP Score in Adolescents With Structural Hyperkyphosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Halic University (Other)
Collaborators: Medipol University (Other); Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HUEK-
Record Dates: First submitted 2021-05-26; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Hyperkyphosis, Adolescent; Scheuermann Disease; Spinal Curvatures
Keywords: Scheuermann Disease; Adolescent Hyperkyphosis; Sagittal Balance; Spinopelvic Parameters
MeSH Terms: conditions — Scheuermann Disease; Spinal Curvatures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to investigate the effect of rıgıd brace treatment on spinopelvic parameters and GAP score in patients with adolescent hyperkyphosis. This was a retrospective analysis of prospectively collected data. Thirty-two patients who were diagnosed with structural hyperkyphosis and treated with CAD-CAM design rigid brace were included in the study in Formed Healthcare Scoliosis Treatment and Brace Center between December 2015-2020.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who diagnosed with Scheuermann's kyphosis or adolescent hyperkyphosis.
* Inıtial curve magnitude between 55-75°
* Patients who followed up at least 6 months
* Patients who wearing CAD-CAM (Computer-Aided Design&Computer-Aided Manufacturing) design TLSO(Thoraco-lumbo-sacral orthosis) kyphosis brace in 16 hours/day or more

Exclusion Criteria:

* History of spinal surgery or trauma
* Patients has kyphosis due to congenital, neuromuscular, traumatic, tumor, infection causes
* Ankylosing spondylitis and other spondyloarthropathies.
* The lack of appropriate full-length lateral radiography with acceptable quality at the baseline or final assessment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 10-18 years patients with Scheuermann's kyphosis or adolescent hyperkyphosis and treated with CAD-CAM design a rigid brace
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-08-16 (Estimated)

PRIMARY OUTCOMES:
Change from kyphosis angle at 6 months | 6 months after from beginning of study
  Change from Baseline kyphosis angle(degree) in standing full-length lateral digital radiographs at 6 months. It will measure between T4-T12 vertebra.
Change from lordosis angle at 6 months | 6 months after from beginning of study
  Change from Baseline lordosis angle(degree) in standing full-length lateral digital radiographs at 6 months. It will measure from the L1-S1 and L4-S1 levels of the vertebra.
Change from the global tilt at 6 months | 6 months after from beginning of study
  Change from Baseline global tilt(degree) in standing full-length lateral digital radiographs at 6 months. The global tilt is the sum of the C7 vertical tilt and the pelvic tilt.
Change from Global Alignment and Proportion (GAP) score at 6 months | 6 months after from beginning
  GAP score is a new pelvic incidence-based proportional method to analyze sagittal alignment and balance, developed by the European Spine Study Group (ESSG). The GAP score evaluates the disproportion, magnitude and distribution of lumbar lordosis, and the global spinopelvic alignment proportionally rather than an absolute numerical value when compared to the ideal calculated for any individual. GAP score has five domains including relative pelvic version, relative lumbar lordosis, lordosis distribution index, relative spinopelvic alignment, and age factor. Scores of each of the four domains vary between 0 to 3 and age factor domain varies between 0 to 1. The total GAP score is between 0 and 13 points and obtained by adding the scores of these five domains. If the total score was 0 to 2, alignment accepted as proportional; 3 to 6 as moderate malalignment; ≥7 was accepted as severe malalignment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen Büyükaslan, PhD(c), Principal Investigator — Medipol University; Kadir Abul, M.D., Study Chair — Başakşehir Çam & Sakura City Hospital; Hürriyet Yılmaz, Prof.Dr., Study Director — Halic University
Locations (1):
- Formed Healthcare Scoliosis Treatment and Brace Center, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No